CLINICAL TRIAL: NCT03645135
Title: Does Goal Elicitation Improve Patient Perceived Involvement?
Brief Title: Does Goal Elicitation Improve Patient Perceived Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 45823
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 1 of 2 study arms arm 1: control arm 2: intervention.
  We will use a random block generator to assign participants to their study arm.
Who Masked: Care Provider
Masking Description: The care provider will not be informed as to which group their patient is in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will be asked to complete a demographics survey and assess their perceived involvement in care after their visit
- Goal elicitation (Experimental): Patients in the intervention group will be asked to list 2 goals for their visit. They will also be asked to complete a demographics survey and access their perceived involvement in care after their visit.
  Interventions: Other: Goal elicitation

INTERVENTIONS:
Other: Goal elicitation — Patients will be asked to list 2 goals for their visit
  Arms: Goal elicitation

SUMMARY:
The purpose of this study is to determine if goal elicitation among orthopaedic patients improves their perceived involvement in care.

DETAILED DESCRIPTION:
This is a RCT with 2 intervention arms. In the first arm, the control arm, patients will be asked to complete a short questionnaire after their visit, to elicit demographic information and perceived involvement in care. The second arm, the intervention arm, will be asked to list 2 goals for their visit and complete a short questionnaire after their visit, to elicit demographic information and perceived involvement in care.

ELIGIBILITY:
Inclusion Criteria:

* New patients visiting the orthopaedic service
* English fluency and literacy

Exclusion Criteria:

* Returning patients
* Children
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Perceived Involvement in Care Scale (PICS) | Immediately after visit
  PICS measures the following: doctor facilitation of patient involvement, level of information exchange, and patient participation in decision making. Scale: 0-13, higher score means higher perceived involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared for this study.